CLINICAL TRIAL: NCT05450133
Title: Relationship Between Systemic Inflammatory Index and Disease Activity in Axial Spondyloarthritis
Brief Title: Hematological Parameters in Axial Spondyloarthritis
Status: Suspended | Type: Observational
Why Stopped: primary researcher is not avaible to recruit participants
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğra İnce, Medical Doctor, Specialist, Bozyaka Training and Research Hospital
Other Study IDs: 2022/PMR_AS
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Disease activity; Inflammatory marker
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- R-ax-Spa: Radiographic axial spondyloarthritis
  Interventions: Other: Systemic inflammatory index; Other: BASDAI; Other: ASDAS-ESR; Other: ASDAS-CRP; Other: MASES
- nR-ax-Spa: Non-radiographic axial spondyloarthritis
  Interventions: Other: Systemic inflammatory index; Other: BASDAI; Other: ASDAS-ESR; Other: ASDAS-CRP; Other: MASES
- Control: Healthy Controls
  Interventions: Other: Systemic inflammatory index

INTERVENTIONS:
Other: Systemic inflammatory index — neutrophil count x platelet count/lymphocyte count
Other: BASDAI — Bath Ankylosing Spondylitis Disease Activity Index includes six questions which includes the following six parameters: fatigue, spinal pain, peripheral joint pain, attachment point inflammation, and duration and severity of morning stiffness. A total score, ranging from 0 to 10, was calculated according to the patients' responses to six questions, with a higher score indicating more severe illness.
  Other Names: Bath Ankylosing Spondylitis Disease Activity Index
  Groups: R-ax-Spa; nR-ax-Spa
Other: ASDAS-ESR — The ASDAS-ESR is deduced using formula that is chosen by the ASAS group. ASDAS-ESR is calculated with the answers of spinal, peripheral pain, morning stiffness on BASDAI, the patient global assessment, and erythrocyte sedimentation rate (mm/h).
  Other Names: Ankylosing Spondylitis Disease Activity Score-ESR
  Groups: R-ax-Spa; nR-ax-Spa
Other: ASDAS-CRP — The ASDAS-CRP is deduced using formula that is chosen by the ASAS group. ASDAS-CRP is calculated with the answers of spinal, peripheral pain, morning stiffness on BASDAI, the patient global assessment, and erythrocyte C-reactive protein (mg/dl).
  Other Names: Ankylosing Spondylitis Disease Activity Score-CRP
  Groups: R-ax-Spa; nR-ax-Spa
Other: MASES — It is used to evaluate the sensitivity of enthesis points by palpation in patients with ankylosing spondylitis. Scoring is done by giving 1 point for sensitive areas and 0 points if there is no sensitivity on the fifth lumbar spinous process, bilateral first and seventh costochondral joints, iliac crystals, posterior and anterior iliac spines, attachment sites of achilles tendon to the calcaneus.
  Other Names: Maastricht Ankylosing Spondylitis Entheses Score
  Groups: R-ax-Spa; nR-ax-Spa

SUMMARY:
Axial spondyloarthritis is an inflammatory disease characterized by the involvement of the sacroiliac joints and the spine. Disease activity and structural changes are determined by using physical examination, imaging studies, laboratory parameters, and patient-reported indices. Among laboratory studies, Erythrocyte sedimentation rate (ESR) and c-reactive protein (CRP) are the most commonly utilized parameters. However, the level of ESR and CRP are inadequate in demonstrating disease activity and inflammation compared to other diseases. In this study, the investigators aimed to analyze and compare the systemic inflammatory index (SII), which is a hematologic parameter between subjects with radiographic axial spondyloarthritis, non-radiographic axial spondyloarthritis, and healthy controls. Secondarily, the relationship between disease activity and enthesitis score and SII scores in patients with radiographic and non-radiographic axial spondyloarthritis will be investigated.

DETAILED DESCRIPTION:
Axial spondyloarthritis is an inflammatory disease characterized by the involvement of the sacroiliac joints and the spine. Disease activity and structural changes are determined by using physical examination, imaging studies, laboratory parameters, and patient-reported indices. Among laboratory studies, Erythrocyte sedimentation rate (ESR) and c-reactive protein (CRP) are the most commonly utilized parameters. ESR and CRP are within the normal range in 40-50% of patients with spondyloarthritis and may remain within the normal range even during active disease. Therefore, the use of biomarkers suitable for the pathophysiology of the disease have been recommended. However, these tests are difficult to access and there is no consensus on showing disease activity. Systemic inflammatory index (SII) is a novel hematologic parameter and previous studies reported the relationship with disease activity in rheumatologic diseases, but the results are inconsistent.

This study will compare the SII between subjects with radiographic and non-radiographic axial spondyloarthritis with healthy subjects. Secondly, the study will investigate the relationship between SII, a new inflammation parameter, and disease activity in patients diagnosed with radiographic and non-radiographic axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with axial spondyloarthritis according to the ASAS classification criteria

Exclusion Criteria:

* Acute/chronic infections
* Presence of other autoimmune diseases
* Diabetes mellitus
* Coronary arterial disease
* Hypertension
* Malignancy
* Hematological diseases
* Liver diseases
* Pregnancy/Lactation
* Renal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Radiographic and non-radiographic axial spondyloarthritis subjects and healthy volunteers will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammatory index | Baseline
  neutrophils * platelets/lymphocytes

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline
  The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
Ankylosing Spondylitis Disease Activity Score (ASDAS)-ESR | Baseline
  <1.3 between "inactive disease" and "low disease activity", <2.1 between "moderate disease activity" and "high disease activity", and >3.5 between "high disease activity" and "very high disease activity".
Ankylosing Spondylitis Disease Activity Score (ASDAS)-CRP | Baseline
  <1.3 between "inactive disease" and "low disease activity", <2.1 between "moderate disease activity" and "high disease activity", and >3.5 between "high disease activity" and "very high disease activity".
Maastricht Ankylosing Spondylitis Entheses Score (MASES) | Baseline
  Maastricht Ankylosing Spondylitis Entheses Score MASES ranging from 0 (0 sites with tenderness) to 13 (worst possible score; 13 sites with tenderness). Negative values indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bugra Ince, Principal Investigator — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Seniz Akcay, Study Director — University of Health Sciences Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Research and Training Hostpital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided by the researchers.

REFERENCES:
- [Background] Song GG, Lee YH. Red cell distribution width, platelet-to-lymphocyte ratio, and mean platelet volume in ankylosing spondylitis and their correlations with inflammation: A meta-analysis. Mod Rheumatol. 2020 Sep;30(5):894-899. doi: 10.1080/14397595.2019.1645373. Epub 2019 Aug 1. PMID 31313609
- [Background] Sezgin M, Tecer D, Kanik A, Kekik FS, Yesildal E, Akaslan E, Yildirim G, Sahin G. Serum RDW and MPV in Ankylosing Spondylitis: Can they show the disease activity? Clin Hemorheol Microcirc. 2017;65(1):1-10. doi: 10.3233/CH-162067. PMID 27258203
- [Background] Malaviya AN, Kalyani A, Rawat R, Gogia SB. Comparison of patients with ankylosing spondylitis (AS) and non-radiographic axial spondyloarthritis (nr-axSpA) from a single rheumatology clinic in New Delhi. Int J Rheum Dis. 2015 Sep;18(7):736-41. doi: 10.1111/1756-185X.12579. Epub 2015 Jul 14. PMID 26172961
- [Background] Tanacan E, Dincer D, Erdogan FG, Gurler A. A cutoff value for the Systemic Immune-Inflammation Index in determining activity of Behcet disease. Clin Exp Dermatol. 2021 Mar;46(2):286-291. doi: 10.1111/ced.14432. Epub 2020 Oct 10. PMID 32869876
- [Background] Wu J, Yan L, Chai K. Systemic immune-inflammation index is associated with disease activity in patients with ankylosing spondylitis. J Clin Lab Anal. 2021 Sep;35(9):e23964. doi: 10.1002/jcla.23964. Epub 2021 Aug 21. PMID 34418163